CLINICAL TRIAL: NCT01366209
Title: A Randomized, Double-Blind, Placebo Controlled, Phase 3 Study of the Efficacy and Safety of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis (ASCEND Trial)
Brief Title: Efficacy and Safety of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: ASCEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIPF-016
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pirfenidone; ASCEND; IPF; FVC
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Arm (Active Comparator)
  Interventions: Drug: Pirfenidone
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone, total daily dose of 2403 mg/ day, given as 3 divided doses 3 times per day.
  Arms: Active Arm
Drug: Placebo — Placebo equivalent given as 3 divided doses 3 times per day.
  Arms: Placebo Arm

SUMMARY:
PIPF-016 (ASCEND) is a Randomized, Double-Blind, Placebo Controlled, Phase 3 Study of the Efficacy and Safety of Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis. The study objectives are to confirm the treatment effect of pirfenidone compared with placebo on change in percent predicted forced vital capacity (%FVC) in patients with idiopathic pulmonary fibrosis (IPF), and to confirm the safety of treatment with pirfenidone compared with placebo in patients with IPF.

ELIGIBILITY:
Select Inclusion Criteria:

1. Diagnosis of idiopathic pulmonary fibrosis (IPF), consistent with the ATS 2011 Guidelines, of 6-48 months' duration
2. Age 40 to 80 at randomization
3. Percent Forced Vital Capacity (%FVC) ≥50% and ≤90% at screening
4. Percent Carbon Monoxide Diffusing Capacity (%DLCO) ≥30% and ≤90% at screening

Select Exclusion Criteria:

1. Forced expiratory volume in one second (FEV1)/FVC ratio <0.8 after administration of bronchodilator at Screening
2. Expected to receive a lung transplant within 1 year from randomization or, for patients at sites in the United States, on a lung transplant waiting list at randomization
3. Known explanation for interstitial lung disease
4. History of asthma or chronic obstructive pulmonary disease
5. Active infection
6. Ongoing IPF treatments including investigational therapy, immunosuppressants, and cytokine modulating agents
7. History of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2011-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: For additional information, call InterMune Medical Information Telephone: 1-888-486-6411, Study Chair — InterMune
Locations (1):
- InterMune Inc., Brisbane, California, United States

REFERENCES:
- [Derived] Kulkarni T, Newton CA, Gupta S, Samara K, Bernstein EJ. The Impact of Autoantibodies on Outcomes in Patients with Idiopathic Pulmonary Fibrosis: Post-Hoc Analyses of the Phase III ASCEND Trial. Pulm Ther. 2024 Sep;10(3):331-346. doi: 10.1007/s41030-024-00267-x. Epub 2024 Jul 29. PMID 39073523
- [Derived] Behr J, Nathan SD, Costabel U, Albera C, Wuyts WA, Glassberg MK, Haller H Jr, Alvaro G, Gilberg F, Samara K, Lancaster L. Efficacy and Safety of Pirfenidone in Advanced Versus Non-Advanced Idiopathic Pulmonary Fibrosis: Post-Hoc Analysis of Six Clinical Studies. Adv Ther. 2023 Sep;40(9):3937-3955. doi: 10.1007/s12325-023-02565-3. Epub 2023 Jun 30. PMID 37391667
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Kreuter M, Lee JS, Tzouvelekis A, Oldham JM, Molyneaux PL, Weycker D, Atwood M, Kirchgaessler KU, Maher TM. Monocyte Count as a Prognostic Biomarker in Patients with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2021 Jul 1;204(1):74-81. doi: 10.1164/rccm.202003-0669OC. PMID 33434107
- [Derived] Glassberg MK, Nathan SD, Lin CY, Morgenthien EA, Stauffer JL, Chou W, Noble PW. Cardiovascular Risks, Bleeding Risks, and Clinical Events from 3 Phase III Trials of Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis. Adv Ther. 2019 Oct;36(10):2910-2926. doi: 10.1007/s12325-019-01052-y. Epub 2019 Aug 10. PMID 31401786
- [Derived] Nathan SD, Costabel U, Albera C, Behr J, Wuyts WA, Kirchgaessler KU, Stauffer JL, Morgenthien E, Chou W, Limb SL, Noble PW. Pirfenidone in patients with idiopathic pulmonary fibrosis and more advanced lung function impairment. Respir Med. 2019 Jul;153:44-51. doi: 10.1016/j.rmed.2019.04.016. Epub 2019 Apr 24. PMID 31153107
- [Derived] Kreuter M, Lederer DJ, Molina-Molina M, Noth I, Valenzuela C, Frankenstein L, Weycker D, Atwood M, Kirchgaessler KU, Cottin V. Association of Angiotensin Modulators With the Course of Idiopathic Pulmonary Fibrosis. Chest. 2019 Oct;156(4):706-714. doi: 10.1016/j.chest.2019.04.015. Epub 2019 Apr 29. PMID 31047956
- [Derived] Nathan SD, Costabel U, Glaspole I, Glassberg MK, Lancaster LH, Lederer DJ, Pereira CA, Trzaskoma B, Morgenthien EA, Limb SL, Wells AU. Efficacy of Pirfenidone in the Context of Multiple Disease Progression Events in Patients With Idiopathic Pulmonary Fibrosis. Chest. 2019 Apr;155(4):712-719. doi: 10.1016/j.chest.2018.11.008. Epub 2018 Nov 22. PMID 30472023
- [Derived] Nathan SD, Lancaster LH, Albera C, Glassberg MK, Swigris JJ, Gilberg F, Kirchgaessler KU, Limb SL, Petzinger U, Noble PW. Dose modification and dose intensity during treatment with pirfenidone: analysis of pooled data from three multinational phase III trials. BMJ Open Respir Res. 2018 Aug 2;5(1):e000323. doi: 10.1136/bmjresp-2018-000323. eCollection 2018. PMID 30116539
- [Derived] Neighbors M, Cabanski CR, Ramalingam TR, Sheng XR, Tew GW, Gu C, Jia G, Peng K, Ray JM, Ley B, Wolters PJ, Collard HR, Arron JR. Prognostic and predictive biomarkers for patients with idiopathic pulmonary fibrosis treated with pirfenidone: post-hoc assessment of the CAPACITY and ASCEND trials. Lancet Respir Med. 2018 Aug;6(8):615-626. doi: 10.1016/S2213-2600(18)30185-1. Epub 2018 Jun 29. PMID 30072107
- [Derived] Paterniti MO, Bi Y, Rekic D, Wang Y, Karimi-Shah BA, Chowdhury BA. Acute Exacerbation and Decline in Forced Vital Capacity Are Associated with Increased Mortality in Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2017 Sep;14(9):1395-1402. doi: 10.1513/AnnalsATS.201606-458OC. PMID 28388260
- [Derived] Kreuter M, Bonella F, Maher TM, Costabel U, Spagnolo P, Weycker D, Kirchgaessler KU, Kolb M. Effect of statins on disease-related outcomes in patients with idiopathic pulmonary fibrosis. Thorax. 2017 Feb;72(2):148-153. doi: 10.1136/thoraxjnl-2016-208819. Epub 2016 Oct 5. PMID 27708114
- [Derived] Nathan SD, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, Glasscock KF, King TE Jr, Lancaster L, Lederer DJ, Lin Z, Pereira CA, Swigris JJ, Valeyre D, Noble PW, Wells AU. Effect of continued treatment with pirfenidone following clinically meaningful declines in forced vital capacity: analysis of data from three phase 3 trials in patients with idiopathic pulmonary fibrosis. Thorax. 2016 May;71(5):429-35. doi: 10.1136/thoraxjnl-2015-207011. Epub 2016 Mar 11. PMID 26968970
- [Derived] Lancaster L, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, King TE Jr, Lederer DJ, Lin Z, Nathan SD, Pereira CA, Swigris JJ, Valeyre D, Noble PW. Safety of pirfenidone in patients with idiopathic pulmonary fibrosis: integrated analysis of cumulative data from 5 clinical trials. BMJ Open Respir Res. 2016 Jan 12;3(1):e000105. doi: 10.1136/bmjresp-2015-000105. eCollection 2016. PMID 26835133
- [Derived] Wijsenbeek MS, Grutters JC, Wuyts WA. Early Experience of Pirfenidone in Daily Clinical Practice in Belgium and The Netherlands: a Retrospective Cohort Analysis. Adv Ther. 2015 Jul;32(7):691-704. doi: 10.1007/s12325-015-0225-1. Epub 2015 Jul 15. PMID 26173796
- [Derived] Lederer DJ, Bradford WZ, Fagan EA, Glaspole I, Glassberg MK, Glasscock KF, Kardatzke D, King TE Jr, Lancaster LH, Nathan SD, Pereira CA, Sahn SA, Swigris JJ, Noble PW. Sensitivity Analyses of the Change in FVC in a Phase 3 Trial of Pirfenidone for Idiopathic Pulmonary Fibrosis. Chest. 2015 Jul;148(1):196-201. doi: 10.1378/chest.14-2817. PMID 25856121
- [Derived] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Arm | Placebo Arm
Started | 278 | 277
Completed | 243 (Participants completing study assessment at Week 52 were completers, even if treatment was withdrawn) | 241
Not Completed | 35 | 36
Not completed — Adverse Event | 6 | 7
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Death | 12 | 19
Not completed — Lung transplantation | 6 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Sponsors decision | 0 | 1
Not completed — Withdrew consent | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Placebo Arm | Total
Number analyzed (Participants) | 278 | 277 | 555
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 88 | 161
  >=65 years | 205 | 189 | 394
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 64 | 120
  Male | 222 | 213 | 435
Region of Enrollment [Number; unit: participants]
  United States | 187 | 184 | 371
  Australia | 33 | 31 | 64
  Brazil | 15 | 16 | 31
  Croatia | 1 | 1 | 2
  Israel | 11 | 9 | 20
  Mexico | 12 | 5 | 17
  New Zealand | 1 | 3 | 4
  Peru | 18 | 26 | 44
  Singapore | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Predicted Forced Vital Capacity (%FVC) From Baseline to Week 52
Time Frame: 52 weeks
Population: Intent to Treat all randomized Patient
Measure: Number; unit: percentage of patients
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 278 | 277
percentage of patients
  Decline or >=10% or Death | 16.5 | 31.8
  No Decline (Change >0%) | 22.7 | 9.7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Active Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 55/278 | 69/277
Other Adverse Events (participants affected / at risk) | 271/278 | 253/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=278) | Placebo Arm (N=277)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (2) | 1 (1)
Angina Pectoris (Cardiac disorders) | 3 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cor Pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratiory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 11 (11) | 14 (16)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intercranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 27 (32)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=278) | Placebo Arm (N=277)
Abdominal pain upper (Gastrointestinal disorders) | 20 (33) | 12 (14)
Constipation (Gastrointestinal disorders) | 32 (38) | 38 (39)
Diarrhoea (Gastrointestinal disorders) | 62 (112) | 60 (101)
Dyspepsia (Gastrointestinal disorders) | 49 (61) | 17 (22)
Flatulence (Gastrointestinal disorders) | 12 (13) | 17 (18)
Gastrooesophageal Reflux (Gastrointestinal disorders) | 33 (36) | 18 (21)
Nausea (Gastrointestinal disorders) | 100 (138) | 37 (46)
Stomach Discomfort (Gastrointestinal disorders) | 24 (38) | 12 (15)
Vomiting (Gastrointestinal disorders) | 36 (74) | 24 (28)
Asthenia (General disorders) | 16 (17) | 11 (12)
Oedema peripheral (General disorders) | 9 (9) | 23 (24)
Pyrexia (General disorders) | 6 (7) | 17 (20)
Bronchitis (Infections and infestations) | 38 (50) | 34 (49)
Influenza (Infections and infestations) | 14 (16) | 12 (12)
Lower respiratory tract infection (Infections and infestations) | 11 (13) | 19 (23)
Nasopharyngitis (Infections and infestations) | 33 (45) | 30 (40)
Sinusitis (Infections and infestations) | 20 (25) | 24 (32)
Upper respiratory tract infection (Infections and infestations) | 61 (78) | 56 (79)
Weight decreased (Investigations) | 35 (35) | 22 (23)
Anorexia (Metabolism and nutrition disorders) | 44 (47) | 18 (19)
Decreased appetite (Metabolism and nutrition disorders) | 20 (23) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (36) | 20 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (35) | 37 (42)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 9 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (18) | 16 (18)
Dizziness (Nervous system disorders) | 49 (88) | 36 (43)
Dysgeusia (Nervous system disorders) | 25 (26) | 11 (12)
Headache (Nervous system disorders) | 72 (117) | 64 (96)
Anxiety (Psychiatric disorders) | 8 (8) | 14 (14)
Depression (Psychiatric disorders) | 9 (9) | 14 (14)
Insomnia (Psychiatric disorders) | 31 (33) | 18 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 70 (104) | 82 (97)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (49) | 49 (66)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 32 (43)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 20 (21)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 14 (14)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 16 (25) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 27 (35) | 19 (20)
Rash (Skin and subcutaneous tissue disorders) | 78 (123) | 24 (27)
Fatigue (General disorders) | 58 (93) | 48 (55)
Urinary tract infection (Infections and infestations) | 8 (12) | 17 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No